CLINICAL TRIAL: NCT02471040
Title: Impact of Recurrent Hypoglycemia on Brain Ketone Metabolism in Type 1 Diabetes
Brief Title: Brain Ketone Metabolism in Type 1 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: 1208010648; 2R01DK101984-06 (NIH)
Record Dates: First submitted 2015-05-28; First posted 2015-06-12 (Estimated); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Type 1 Diabetes; Hypoglycemia
Keywords: brain metabolism; cognitive function
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hypoglycemia | interventions — 3-Hydroxybutyric Acid; Saline Solution; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: The added 3rd arm does not apply to the crossover design.
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Type 1 diabetic subjects (Experimental): Subjects will undergo a hyperinsulinemic-hypoglycemic clamp with a target glucose level of 55mg/dl. Once a stable glycemic state is reached, subjects will receive a bolus-continuous infusion beta-hydroxybutyrate (BHB) or infusion of a comparable volume of normal saline (placebo) to control for possible volume effects for the remainder of the study. Throughout the BHB or saline infusion cognitive function will be tested via a standardized testing battery.
  Interventions: Drug: Beta-hydroxybutyrate; Other: Normal Saline
- Healthy Subjects (Active Comparator): Healthy control subjects will undergo a hyperinsulinemic-hypoglycemic clamp with a target glucose level of 55mg/dl. Once a stable glycemic state is reached, subjects will receive a bolus-continuous infusion beta-hydroxybutyrate (BHB) or infusion of a comparable volume of normal saline (placebo) to control for possible volume effects for the remainder of the study. Throughout the BHB or saline infusion cognitive function will be tested via a standardized testing battery.
  Interventions: Drug: Beta-hydroxybutyrate; Other: Normal Saline
- Healthy Subjects CONTROL (Active Comparator): Healthy control subjects will undergo a hyperinsulinemic-hypoglycemic clamp with a target glucose level of 55mg/dl. Once a stable glycemic state is reached, subjects will undergo an NMR test to characterize brain metabolism under hypoglycemia.
  Interventions: Other: Normal Saline

INTERVENTIONS:
Drug: Beta-hydroxybutyrate — Both healthy subjects and type 1 diabetic subjects will receive a bolus-continuous infusion of 40umol/min/kg of BHB for 5 min, followed by a 12µmol/min/kg of BHB or infusion of a comparable volume of normal saline (placebo) to control for possible volume effects for the remainder of the study.
  Other Names: BHB
  Arms: Healthy Subjects; Type 1 diabetic subjects
Other: Normal Saline — Both healthy subjects and type 1 diabetic subjects will receive a bolus-continuous infusion of 40umol/min/kg of BHB for 5 min, followed by a 12µmol/min/kg of BHB or infusion of a comparable volume of normal saline (placebo) to control for possible volume effects for the remainder of the study.
  Other Names: NaCl 0.9%

SUMMARY:
This study is designed to examine the value of infusing BHB in type 1 diabetic subjects during experimentally induced hypoglycemic episode in conjunction with testing of cognitive function. This will lay the basis for subsequent trials exploring the novel use of therapeutic doses of oral ketone formulations that are currently under commercial development, which could serve as adjunct therapies to protect the brain from hypoglycemia in type 1 diabetic subjects experiencing recurrent hypoglycemia.

DETAILED DESCRIPTION:
Healthy controls as well as type 1 diabetic subjects will undergo a hyperinsulinemic-hypoglycemic clamp with concomitant BHB or saline (control) infusion in random order. During each experimental condition the participants will complete a battery of validated cognitive tests that are sensitive to the cognitive impairment typically caused by hypoglycemia. An additional healthy control arm was added to the study design after the initial registration as a 2 arm study, to provide imaging results of normal healthy responses to hypoglycemia.

ELIGIBILITY:
Inclusion Criteria:

1. Type 1 diabetes mellitus of > 5 years (C-peptide negative, age 18-60 years, on intensive insulin therapy (HbA1c <7.5%)
2. Non-diabetic volunteers, age 18-65 years that do not meet any of the exclusion criteria.

Exclusion Criteria:

1. Pregnancy
2. Significant baseline anemia (hemoglobin <11.0 or hematocrit < 33%)
3. A history of liver cirrhosis or porto-caval shunt surgery.
4. Any contraindications for MRI scanning.
5. Subjects that follow a vegetarian diet
6. Subjects that exercise heavily on a regular basis (i.e. marathon runners, body builders or other forms of excessive exercise as determined by the PI)
7. Subjects with a history of anxiety/ panic attacks

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2013-05-14 (Actual); Primary Completion 2022-04-04 (Actual); Study Completion 2022-04-04 (Actual)

PRIMARY OUTCOMES:
Cognitive Function | Under clamped hypoglycemia (50 min from start)
  Subjects from all groups will be studied using the NIH Toolbox Cognition Battery, which includes measurements of Executive Function, Attention, Episodic Memory, Language, Processing Speed and Working Memory.

CONTACTS AND LOCATIONS:
Overall Officials: Raimund Herzog, MD, Principal Investigator — Yale University
Locations (1):
- Yale New Haven Hospital, New Haven, Connecticut, United States

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-04): https://cdn.clinicaltrials.gov/large-docs/40/NCT02471040/Prot_SAP_000.pdf